CLINICAL TRIAL: NCT01989312
Title: Can we Gain an Advantage by Combining Distal Median, Radial and Ulnar Nerve Blocks With Supraclavicular Block? A Randomized Controlled Study
Brief Title: The Simultaneous Use of Supraclavicular and Distal Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Basak Ceyda MECO, MD,DESA, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 03-99-12
Record Dates: First submitted 2013-10-31; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Orthopaedic Disorders; Nerve Block; Anaesthesia
Keywords: ultrasound; peripheral nerves; anesthetics; local
MeSH Terms: interventions — Lidocaine; Epinephrine; Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- supraclavicular block (Active Comparator): A supraclavicular block with 32 mL of lidocaine 1.5% + epinephrine 5µg/mL was performed for the anaesthetic management of the forearm and hand.
  Interventions: Procedure: intravenous cannulation.; Device: Intravenous cannulation.; Device: Routine ASA monitoring; Drug: Premedication midazolam; Drug: Lidocaine; Drug: Epinephrine
- Supraclavicular and median, ulnar, radial blocks (Active Comparator): Patients in this group received 20 mL of lidocaine 1.5% + epinephrine 5µg/mL for supraclavicular block and after the supraclavicular block they recieved a distal median, radial, and ulnar nerve blocks using 50:50 mixture of lidocaine 2% + levobupivacaine 0.5% (4 mL/nerve).
  Interventions: Procedure: Supraclavicular block and ultrasound-guided ulnar, median and radial nerve blocks.; Device: Intravenous cannulation.; Device: Routine ASA monitoring; Drug: Premedication midazolam; Drug: Lidocaine; Drug: Epinephrine; Drug: Levobupivacaine

INTERVENTIONS:
Procedure: intravenous cannulation. — A 18-or 20-gauge intravenous (iv) catheter was placed to the contralateral arm according to the surgical site
  Arms: supraclavicular block
Procedure: Supraclavicular block and ultrasound-guided ulnar, median and radial nerve blocks. — Supraclavicular block with 20 mL of lidocaine 1.5% + epinephrine 5µg/mL and the addition of ultrasound-guided ulnar, median and radial nerve blocks. For that 12 mL of local anesthetic solution of a 50:50 mixture of lidocaine 2% and levobupivacaine 0.5% (4 mL/nerve) was used.
  Arms: Supraclavicular and median, ulnar, radial blocks
Device: Intravenous cannulation. — A 18-or 20-gauge intravenous (iv) catheter was placed to the contralateral arm according to the surgical site
Device: Routine ASA monitoring — Monitorization with ECG, noninvasive blood pressure and spO2.
Drug: Premedication midazolam — Premedication with 0.03 mg/kg midazolam iv
Drug: Lidocaine
Drug: Epinephrine
Drug: Levobupivacaine
  Arms: Supraclavicular and median, ulnar, radial blocks

SUMMARY:
The aim of this study is to compare the combined ultrasound-guided supraclavicular brachial plexus block and distal median, radial, and ulnar nerve blocks, with supraclavicular block alone.

Sixty two patients undergoing upper extremity surgery will be randomized to supraclavicular only (Group S, n=31) or supraclavicular + distal (Group SD, n=31) group. Patients in group S will receive 32 mL of lidocaine 1.5% + epinephrine 5µg/mL and in group SD receive 20 mL of lidocaine 1.5% + epinephrine 5µg/mL followed by a distal median, radial, and ulnar nerve blocks using 50:50 mixture of lidocaine 2% + levobupivacaine 0.5% (4 mL/nerve). Sensory and motor block of the ulnar, median, radial and musculocutaneous nerves will be assessed every 5 minutes starting at the 10th minutes. The imaging, needling and performance times will be recorded. Also the onset and anesthesia related times, need for analgesic and first analgesic time will be noted.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 80 years old patient
* American Society of Anesthesiologists (ASA) physical status I-III
* Scheduled for elective hand and forearm surgery

Exclusion Criteria:

* patient refusal
* preexisting neuropathy
* coagulopathy
* allergy to agents used
* pregnancy
* body mass index > 35 kg/m2
* chronic obstructive pulmonary disease
* infection or previous surgery in the supraclavicular area
* systemic infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The time required after a supraclavicular block alone or a supraclavicular block combined with distal blocks, to achieve a sensory and motor block needed for surgery. | All patients will be followed up during the block procedure and during the surgery. Also, after the surgery patients will be followed up to 7 days postoperatively.
  The onset time of supraclavicular plexus block and the onset time of supraclavicular block combined with distal median, radial, and ulnar nerve blocks will be followed up. The time needed to achieve a surgical block will be assessed in both groups. The difference between the 2 groups will be compared and analysed. For this an investigator blinded to the group allocation will evaluate the sensorial pinprick and motor blocks of the ulnar, median, radial and musculocutaneous nerves every 5 minutes starting at the 10th minutes until 30th minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Ceyda Meco, MD, DESA, Principal Investigator — Ankara University Faculty of Medicine
Locations (1):
- Ankara University Faculty of Medicine, Ibni Sina Hospital colonoscopy lab, Ankara, Turkey (Türkiye)